CLINICAL TRIAL: NCT01392911
Title: A Phase IIA Dose Ranging Trial to Evaluate the Safety, Tolerability, Extended Early Bactericidal Activity and Pharmacokinetics of Higher Doses of Rifampicin in Adult Subjects With Newly Diagnosed, Uncomplicated, Smear-Positive, Pulmonary Tuberculosis
Brief Title: Safety, Tolerability, Extended Early Bactericidal Activity and PK of Higher Doses Rifampicin in Adults With Pulmonary TB
Acronym: HR1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Department of Clinical Pharmacy, University Medical Centre St Radboud, The Netherlands. (Other); University Centre for Chronic Diseases Dekkerswald, Groesbeek, NL (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PanACEA - RUNMC - HR1; 2007.23011.01 (Other Grant/Funding Number: EDCTP - Boeree.PanACEA_IP)
Record Dates: First submitted 2011-06-14; First posted 2011-07-13 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Tuberculosis (TB)
Keywords: Dose Ranging; Extended Early Bactericidal Activity; Maximum tolerable dose; Pharmacokinetics; Pulmonary Tuberculosis; Rifampicin; Rifafour; Safety; Tolerability; Max Tolerable Dose
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 10 mg/kg rifampicin (Active Comparator): 7 Days monotherapy with 10 mg/kg rifampicin followed by 7 days standard TB treatment, i.e. Rifafour® e275 once daily including the standard dose of rifampicin.
  Interventions: Drug: Rifampicin
- 20 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 20 mg/kg rifampicin followed by 7 days combination therapy consisting of 20 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 25 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 25 mg/kg rifampicin followed by 7 days combination therapy consisting of 25 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 30 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 30 mg/kg rifampicin followed by 7 days combination therapy consisting of 30 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 35 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 35 mg/kg rifampicin followed by 7 days combination therapy consisting of 35 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 40 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 40 mg/kg rifampicin followed by 7 days combination therapy consisting of 40 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 45 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 45 mg/kg rifampicin followed by 7 days combination therapy consisting of 45mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 50 mg/kg rifampicin (Experimental): 7 Days monotherapy with 50 mg/kg rifampicin followed by 7 days combination therapy consisting of 50 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin
- 55 mg/kg Rifampicin (Experimental): 7 Days monotherapy with 55 mg/kg rifampicin followed by 7 days combination therapy consisting of 55 mg/kg rifampicin plus the standard doses of isoniazid, ethambutol and pyrazinamide.
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Rifampicin — High dose rifampicin
  Other Names: Rifadin; Rifafour

SUMMARY:
This is the first trial in a series of clinical trials that aim to bring the concept of high dose rifampicin beyond phase II of clinical development.

The safety, tolerability, extended early bactericidal activity (EBA) and pharmacokinetics of several doses of Rifampicin with or without standard doses of Isoniazid, Pyrazinamide and Ethambutol in adults with newly diagnosed, uncomplicated, smear positive, pulmonary TB will be assessed. The objective of this study is to find the maximum tolerable dose of Rifampicin as monotherapy and in combination with the currently available Isoniazid, Pyrazinamide and Ethambutol.

The subjects will be in the study for 24-31 days. After a screening period of 9-3 days, the subjects will receive treatment with Rifampicin as single drug during 7 days (monotherapy). This treatment will be followed by treatment with 7 days of Rifampicin and Isoniazid, Pyrazinamide and Ethambutol (combination therapy), and 7-8 days treatment with standard TB medication.

All subjects will be closely monitored for side effects. This monitoring will include daily interviews and physical examination, and ECG evaluation and blood and urine analyses at specific intervals.

During the 7 days of monotherapy, after the second day of the combination therapy and at the end of the combination therapy, overnight sputum will be collected from the patients to investigate the potency of high dose rifampicin to reduce this number of bacilli.

The Rifampicin dose will be increased step by step and group by group. The control group will receive the standard dose of 10 mg Rifampicin/kg, whereas the first treatment group will receive 20 mg/kg. The Rifampicin dose will only be further increased for a next group of patients, if this is expected to be safe.

Rifampicin is widely available and not expensive. Physicians all over the world have experience with this drug and its adverse effects. Should this study be successful, the highest dose of Rifampicin that this safe and tolerable will be given to a larger group of patients. in the next study.

If increasing the dose of Rifampicin proves to be safe and effective, a higher dose of Rifampicin could be implemented broadly and quickly, and it would benefit many patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is able and willing to provide written, informed consent prior to all trial-related procedures including HIV testing.
2. The patient is aged between 18 and 65 years, inclusive.
3. The patient has a body weight (in light clothing and with no shoes) between 40 and 85 kg, inclusive.
4. The patient is a newly diagnosed, previously untreated, uncomplicated, sputum smear-positive, pulmonary TB patient.
5. The patient has a normal chest X-ray or a picture which in the opinion of the Investigator is compatible with TB.
6. The patient is sputum positive on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale (Appendix 4)).
7. The patient is able to produce an adequate volume of sputum as estimated from a spot assessment (estimated 10 ml or more overnight production).
8. The patient has a negative serum pregnancy test (female subjects of childbearing potential only)
9. The patient agrees to use a highly effective method of birth control (i.e. two of the following precautions: tubal ligation, vaginal diaphragm, intrauterine device, condom, oral contraceptives, contraceptive implant, combined hormonal patch, combined injectable contraceptive or depot-medroxyprogesterone acetate, partner(s) has/have had a vasectomy) throughout the participation in the trial and for 1 week after last dose, unless she and her partner(s) are sterile (that is, women who have had a bilateral oophorectomy and/or hysterectomy or have been postmenopausal for at least 12 consecutive months; men who have had bilateral orchidectomy).
10. A Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs).

Exclusion Criteria:

1. The patient is in poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
2. Rifampicin-resistant bacteria have been detected in the patient's sputum specimen collected within the Pre-Treatment Period and tested at the study laboratory.
3. The patient has received treatment with any drug active against MTB within the 3 months prior to Visit 1: isoniazid, ethambutol, amikacin, cycloserine, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, quinolones, thioamides.
4. The patient has a history of allergy to isoniazid, ethambutol, rifampicin and pyrazinamide,
5. The patient has a history of previous TB.
6. The patient has Hepatitis B.
7. The patient had Hepatitis C.
8. The patient is infected with HIV and has a CD4 count < 350 cells/uL (Visit 1).
9. The patient is receiving antiretroviral therapy (ART).
10. The patient has been taking rifampicin within 30 days prior to Visit 1.
11. The patient is a diabetic using insulin.
12. The patient is pregnant or breast-feeding (female patients only).
13. The patient has a history and/or presence (or evidence) of neuropathy or epilepsy.
14. The patient has a history of or current clinically relevant cardiovascular disorder such as:

    1. heart failure, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia or status after myocardial infarction.
    2. family history of sudden death of unknown or cardiac-related cause, or of prolonged QTc interval.
15. Concomitant use of any drug known to prolong QTc interval (including amiodarone, bepridil chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine).
16. The patient has any disease or condition in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug or their components.
17. There is clinically significant evidence of extrathoracic TB (miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
18. Evidence of serious lung conditions other than TB or uncontrolled obstructive bronchial disease.
19. The patient has clinically relevant changes in the ECG such as atrioventricular (AV) block, prolongation of the QRS complex over 120 milliseconds, or of either the QTcF or QTcB interval over 450 milliseconds on the screening ECG.
20. There is any evidence showing that the patient has renal impairment, including but not limited to serum creatinine levels above the upper limit of the laboratory reference range.
21. The patient has abnormal alanine aminotransferase (ALT) and/or aspertate transferase (AST) levels > 1 times the upper limit of the laboratory reference range (at Visit 1).
22. There is evidence showing the patient has clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
23. The patient has any disease or condition in which any of the medicinal products listed in the section pertaining to prohibited medication is used.
24. The patient has a known or suspected, current or history of drug or amphetamine abuse, within the past 2 years, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the patient.
25. The patient has a known or suspected current history of significant alcohol consumption, i.e. more than 20 units/week, within the past 2 years.
26. The patient used any drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes within 30 days prior to Visit 4 (including xenobiotics, quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan). Exceptions may be made for patients who have received 3 days or less of one of these drugs or substances, if there has been a wash-out period prior to Visit 4 equivalent to at least 5 half-lives of that drug or substance.
27. The patient used any therapeutic agents known to alter any major organ function (e.g., barbiturates, phenothiazines, cimetidine) within 14 days prior to Visit 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2011-06; Primary Completion 2018-07 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events associated with increasing doses of rifampicin when administered as a single drug. | 7 days
The incidence and severity of adverse events associated with increasing doses of rifampicin when combined with isoniazid, pyrazinamide and ethambutol. | 7 days

SECONDARY OUTCOMES:
The Early Bactericidal Activity (EBA) expressed as the fall of colony forming units per mL of sputum per day at the intervals: Baseline to Day 2, Baseline to Day 7, Baseline to Day 14, and Day 8 to Day 14. | Visit 2 (Day -2) (if needed also on Visit 3 (Day -1)), Visit 4 (Day 1), Visit 5 (Day 2), Visit 6 (Day 3), Visit 7 (Day 4), Visit 8 (Day 5), Visit 9 (Day 6), Visit 10 (Day 7), Visit 12 (Day 9) and Visit 17 (Day 14)
The change in Time to Positivity (TTP) as measured in the Mycobacterium Growth Indicator Tube (Bactec MGIT960 system) at the intervals: Baseline to Day 2, Baseline to Day 7, Baseline to Day 14, and Day 8 to Day 14. | Visit 2 (Day -2) (if needed also on Visit 3 (Day -1)), Visit 4 (Day 1), Visit 5 (Day 2), Visit 6 (Day 3), Visit 7 (Day 4), Visit 8 (Day 5), Visit 9 (Day 6), Visit 10 (Day 7), Visit 12 (Day 9) and Visit 17 (Day 14)
The area under the plasma concentration versus time curve (AUC) of rifampicin, and if possible also the AUC of pyrazinamide, isoniazid and ethambutol after 7 days of monotherapy with rifampicin and after 7 days of combination therapy | Day 7 and Day 14
Pharmacodynamic endpoints for single dose rifampicin (assessed at Day 7) and or rifampicin, isoniazid, pyrazinamide and ethambutol when administered together (assessed at Day 14). | Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Martin Boeree, MD, PhD, Study Chair — Radboud university medical center, University Centre for Chronic Deseases Dekkerswald; Rob Aarnoutse, PharmD, PhD, Study Chair — Radboud University Medical Center; Andreas Diacon, MD, Principal Investigator — TASK Applied Science; Rodney Dawson, MD, Principal Investigator — University of Cape Town Lung Institute
Locations (2):
- South Africa (2):
  - TASK Applied Science, Bellville
  - University of Cape Town Lung Institute, Mowbray

REFERENCES:
- [Derived] Te Brake LHM, de Jager V, Narunsky K, Vanker N, Svensson EM, Phillips PPJ, Gillespie SH, Heinrich N, Hoelscher M, Dawson R, Diacon AH, Aarnoutse RE, Boeree MJ; PanACEA Consortium. Increased bactericidal activity but dose-limiting intolerability at 50 mg.kg-1 rifampicin. Eur Respir J. 2021 Jul 8;58(1):2000955. doi: 10.1183/13993003.00955-2020. Print 2021 Jul. PMID 33542056
- [Derived] Svensson RJ, Svensson EM, Aarnoutse RE, Diacon AH, Dawson R, Gillespie SH, Moodley M, Boeree MJ, Simonsson USH. Greater Early Bactericidal Activity at Higher Rifampicin Doses Revealed by Modeling and Clinical Trial Simulations. J Infect Dis. 2018 Aug 14;218(6):991-999. doi: 10.1093/infdis/jiy242. PMID 29718390
- [Derived] Boeree MJ, Diacon AH, Dawson R, Narunsky K, du Bois J, Venter A, Phillips PP, Gillespie SH, McHugh TD, Hoelscher M, Heinrich N, Rehal S, van Soolingen D, van Ingen J, Magis-Escurra C, Burger D, Plemper van Balen G, Aarnoutse RE; PanACEA Consortium. A dose-ranging trial to optimize the dose of rifampin in the treatment of tuberculosis. Am J Respir Crit Care Med. 2015 May 1;191(9):1058-65. doi: 10.1164/rccm.201407-1264OC. PMID 25654354